CLINICAL TRIAL: NCT05378997
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study in Healthy Male and Female Volunteers to Investigate the Safety, Tolerability, and Pharmacokinetics of Ascending Topical Doses of TCP-25 Applied to Epidermal Suction Blister Wounds and in Patients With Non-Healing Leg Ulcers and Patients With Dystrophic Epidermolysis Bullosa
Brief Title: Safety, Tolerability, and Pharmacokinetics of Ascending Topical Doses of TCP-25 Applied to Epidermal Suction Blister Wounds, Non-Healing Leg Ulcers and Patients With Dystrophic Epidermolysis Bullosa.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xinnate AB (Industry)
Collaborators: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCP-25-001; 2021-004728-14 (EudraCT Number)
Record Dates: First submitted 2022-04-25; First posted 2022-05-18 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Blister; Wound of Skin; Epidermolysis Bullosa; Varicose Ulcer of Lower Limb
Keywords: acute epidermal wounds; suction blister; healthy volunteers
MeSH Terms: conditions — Blister; Epidermolysis Bullosa

STUDY DESIGN:
Intervention Model Description: Part I: Multiple topical doses of TCP-25 will be administered in 3 sequential dose groups, each of 8 subjects. Within each cohort, the subjects will receive TCP-25 on one wound on each thigh and placebo on one wound on each thigh in a randomized fashion as topical treatment. In Part II: Multiple topical doses of TCP-25 will be administered to 6 patients with non-healing leg ulcers. In Part III: Up to 4 dose levels of TCP-25 will be administered in up to 5 patients with DEB by topical application of TCP-25 gel of two concentrations.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose group 1 (Experimental): 0.15 mL of TCP-25 gel (0.86 mg/mL) or 0.15 mL placebo gel per wound applied as topical treatment on days 1, 2, 3, 5, and 8
  Interventions: Drug: TCP-25 gel 0.86 mg/ml or placebo gel
- Dose group 2 (Experimental): 0.15 mL of TCP-25 gel (2.9 mg/mL) or 0.15 mL placebo gel per wound applied as topical treatment on days 1, 2, 3, 5, and 8
  Interventions: Drug: TCP-25 gel 2.9 mg/ml or placebo gel
- Dose group 3 (Experimental): 0.15 mL of TCP-25 gel (8.6 mg/mL) or 0.15 mL placebo gel per wound applied as topical treatment on days 1, 2, 3, 5, and 8
  Interventions: Drug: TCP-25 gel 8.6 mg/ml or placebo gel

INTERVENTIONS:
Drug: TCP-25 gel 0.86 mg/ml or placebo gel — TCP-25 gel (0.86 mg/mL) applied to two wounds per patient and placebo gel applied to two wounds per patient
  Arms: Dose group 1
Drug: TCP-25 gel 2.9 mg/ml or placebo gel — TCP-25 gel (2.9 mg/mL) applied to two wounds per patient and placebo gel applied to two wounds per patient
  Arms: Dose group 2
Drug: TCP-25 gel 8.6 mg/ml or placebo gel — TCP-25 gel (8.6 mg/mL) applied to two wounds per patient and placebo gel applied to two wounds per patient
  Arms: Dose group 3

SUMMARY:
This is a three-part, Phase I, first-in-human study designed to evaluate the safety, tolerability, and potential systemic exposure of multiple topical doses of TCP-25. Part I includes healthy volunteers with acute epidermal wounds formed by the suction blister technique. Part II includes patients with non-healing leg ulcers and Part III patients with dystrophic epidermolysis bullosa (DEB).

ELIGIBILITY:
Part I:

Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy male or female subject 18-60 years (inclusive) of age at the time of signing the informed consent.
3. Body Mass Index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2.
4. Healthy and intact skin where the blister suction wounds will be induced.
5. Women of childbearing potential (WOCBP) must have a documented negative serum pregnancy test done at the screening visit, within 4 weeks prior to suction blister formation and the start of study treatment.

   WOCBP must practice abstinence (only allowed when this is the preferred and usual lifestyle of the subject) or must agree to use a highly effective method of contraception with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD] or intrauterine hormone-releasing system [IUS]) from at least 4 weeks prior to dose to 4 weeks after last dose. Female subjects must refrain from donating eggs from the date of dosing until 3 months after dosing with the IMP. Their male partner must agree to use a condom during the same time frame if he has not undergone vasectomy.

   Women of non-childbearing potential are defined as pre-menopausal females who are sterilised (tubal ligation or permanent bilateral occlusion of fallopian tubes); or females who have undergone hysterectomy or bilateral oophorectomy; or post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with detection of follicle stimulating hormone [FSH] 25-140 IE/L is confirmatory).

   Male subjects must be willing to use condom or be vasectomised or practice sexual abstinence to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the date of last dosing until 3 months after the last dosing with the IMP. Their female partner of child-bearing potential must use contraceptive methods with a failure rate of < 1% to prevent pregnancy (see above).
6. Clinically relevant medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Disease that may interfere with wound healing, e.g., diabetes type I/II, arterial-, renal-, liver, or cardiac insufficiency, chronic obstructive lung disease, cancer, autoimmune disease, edema at the study site, severe obesity, or previous known wound healing problems, as judged by the investigator.
3. Active skin disease, e.g., dermatitis, psoriasis and wounds, and/or tattoos in the areas where suction blister wounds will be induced, as judged by the investigator.
4. Any planned major surgery within the duration of the study.
5. After 10 minutes supine rest at the time of screening, any vital signs values outside the following ranges:

   * Systolic blood pressure <90 or >160 mmHg, or
   * Diastolic blood pressure <50 or >100 mmHg, or
   * Pulse <40 or >90 beats per minute (bpm)
6. Any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
7. Current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than three times per week is allowed before screening visit.
8. Female subjects who are pregnant or lactating or planning a pregnancy.
9. Systemic immunosuppressive treatment.
10. Subjects who are currently receiving or have received the following treatments within 2 weeks prior to screening are excluded from the study: - systemic corticosteroids or immunosuppressant agents; or - antibiotics via any route
11. Regular use of anticoagulants (i.e., heparin, warfarin, coumarins, other anticoagulants per Investigator's judgement) or non-steroidal anti-inflammatory drugs (NSAIDs) within 2 weeks prior to the (first) administration of IMP, at the discretion of the Investigator.
12. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to TCP-25 or to any excipients of the hydrogel.
13. Planned treatment or treatment with another investigational drug within 3 months prior to Day -1.
14. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
15. Presence or history of drug abuse, as judged by the Investigator
16. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the three months prior to screening.
17. Involvement in the planning and/or conduct of the study.
18. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Part II:

Inclusion criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Male patient, or female patient of non-childbearing potential, ≥40 years of age at the time of signing the informed consent.
3. Male subjects must be willing to use condom or be vasectomized or practice sexual abstinence to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the date of last dosing until 3 months after the last dosing with the IMP. Their female partner of child-bearing potential must use contraceptive methods with a failure rate of < 1% to prevent pregnancy.

   Women of non-childbearing potential are defined as pre-menopausal females who are sterilised (tubal ligation or permanent bilateral occlusion of fallopian tubes); or females who have undergone hysterectomy or bilateral oophorectomy; or post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with detection of follicle stimulating hormone [FSH] 25-140 IU/L is confirmatory).
4. Clinically relevant medical history, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.
5. Patients diagnosed with venous insufficiency by relevant physiological tests including doppler or venous plethysmography or diagnosed by relevant clinical evaluations.
6. Systolic index > 0.6 (Data from medical records from the last 2 years, or the assessment should be repeated at the screening visit).
7. Ulcer duration > 6 weeks
8. Total target ulcer area applicable for treatment: ≤ 30 cm2 (as measured with the Silhouette imaging equipment at the screening visit). (The target ulcer area may not consist of >2 separate ulcers.)
9. Ability to tolerate compression bandaging.
10. Willing to attend study site visits.

Exclusion criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Disease that may interfere with wound healing, e.g., diabetes type I/II, arterial-, renal-, liver, or cardiac insufficiency, chronic obstructive lung disease, cancer, autoimmune disease, edema at the study site, severe obesity, or previous known wound healing problems, as judged by the Investigator.
3. Active skin disease, e.g., dermatitis, psoriasis and wounds, and/or tattoos in the areas where suction blister wounds will be induced, as judged by the Investigator.
4. Any planned major surgery within the duration of the study.
5. After 10 minutes supine rest at the time of screening, any vital signs values outside the following ranges:

   * Systolic blood pressure <90 or >160 mmHg, or
   * Diastolic blood pressure <50 or >100 mmHg, or
   * Pulse <40 or >90 beats per minute (bpm)
6. Any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
7. Current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than three times per week is allowed before screening visit.
8. Female subjects who are pregnant or lactating or planning a pregnancy.
9. Systemic immunosuppressive treatment.
10. Subjects who are currently receiving or have received the following treatments within 2 weeks prior to screening are excluded from the study:

    * systemic corticosteroids or immunosuppressant agents; or
    * antibiotics via any route
11. Regular use of anticoagulants (i.e., heparin, warfarin, coumarins, other anticoagulants per Investigator's judgement) or non-steroidal anti-inflammatory drugs (NSAIDs) within 2 weeks prior to the (first) administration of IMP, at the discretion of the Investigator.
12. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to TCP-25 or to any excipients of the hydrogel.
13. Planned treatment or treatment with another investigational drug within 3 months prior to Day -1.
14. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
15. Presence or history of drug abuse, as judged by the Investigator.
16. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the three months prior to screening.
17. Involvement in the planning and/or conduct of the study.
18. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

9.5.2 Part II: Exclusion criteria

Patients must not enter the study if any of the following exclusion criteria are fulfilled:

1. Presence or documented illness, which in the Investigator's opinion may negatively affect wound healing or interfere with the study conduct.
2. Target wound present for more than 5 years.
3. Clinical signs of infection in or around the wound in need of antibiotic treatment.
4. Albumin <25 g/L or capillary Hb <90 g/L, or HbA1c > 70 mmol/mol at the time of the screening visit.
5. Any planned major surgery within the duration of the study.
6. Patients who are currently receiving or have received the following treatments within 2 weeks prior to screening are excluded from the study:

   * systemic corticosteroids above 5 mg prednisolone or equivalent, or
   * immunosuppressant agents; or
   * antibiotics via any route.
7. Regular use of anticoagulants (i.e., heparin, warfarin, coumarins, other anticoagulants affecting APTT and/or PK/INR per Investigator's judgement) within 2 weeks prior to the (first) administration of IMP, at the discretion of the Investigator.
8. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to TCP-25 or to any excipients of the hydrogel.
9. Planned treatment or treatment with another investigational drug within 3 months prior to Day -1.
10. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the three months prior to screening.
11. Involvement in the planning and/or conduct of the study.
12. Investigator considers the patient unlikely to comply with study procedures, restrictions and requirements.

Part III:

Inclusion criteria:

1. Willing and able to give written informed consent for participation in the study. For 15 to 17-year-olds: A separate consent is required from both (if applicable) the patient's parents/legal guardians.
2. Male or female patient with documented diagnosis of inherited DEB, ≥15 years of age at the time of signing the informed consent.
3. Male patients must be willing to use condom or be vasectomized or practice sexual abstinence to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the date of last dosing until 3 months after the last dosing with the IMP. Their female partner of child-bearing potential must use contraceptive methods with a failure rate of < 1% to prevent pregnancy.

   WOCBP must practice abstinence (only allowed when this is the preferred and usual lifestyle of the patient) or must agree to use a highly effective method of contraception with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD] or intrauterine hormone-releasing system [IUS]) from at least 4 weeks prior to dose to 4 weeks after last dose. Female patients must refrain from donating eggs from the date of dosing until 3 months after dosing with the IMP. Their male partner must agree to use a condom during the same time frame if he has not undergone vasectomy.

   Women of non-childbearing potential are defined as pre-menopausal females who are sterilised (tubal ligation or permanent bilateral occlusion of fallopian tubes); or females who have undergone hysterectomy or bilateral oophorectomy; or post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with detection of follicle stimulating hormone [FSH] 25-140 IU/L is confirmatory).
4. Clinically relevant medical history at the time of screening, as judged by the Investigator.
5. Presence of two target wound areas of 50 cm2. The primary wound area should not be located at anatomical sites with high likelihood of accidental trauma (e.g., knee, elbow). The secondary wound area could be located at anatomical sites with high likelihood of accidental trauma or be within the higher age span. Both wound areas should meet all the following characteristics:

   1. Including open wound with a surface area of ≤ 30 cm2 (as measured with the Silhouette imaging equipment at the screening visit).
   2. At Visit 2 (first IMP treatment), each target wound should not present a surface reduction ≥ 30 % from the Screening visit.
   3. Wound aged ≥ 3 weeks to < 9 months at the Screening visit.
6. Presence of a reference wound area of 50 cm2 to be treated with standard of care only and to be included in the exploratory assessment. The wound area should match the primary wound area for following characteristics:

   1. Including open wound with a surface area of ≤ 30 cm2 (as measured with the Silhouette imaging equipment at the screening visit).
   2. At Visit 2 (first IMP treatment), the wound should not present a surface reduction ≥ 30 % from the Screening visit.
   3. Wound aged ≥ 3 weeks to < 9 months at the Screening visit.
   4. Not located at anatomical sites with high likelihood of accidental trauma (e.g., knee, elbow).
7. Willing to attend study site visits.

Exclusion criteria

1. Any subtype of EB other than DEB.
2. EB index wounds that have infection in need of systemic antibiotic treatment.
3. Presence of or documented illness, which in the Investigator's opinion may negatively affect wound healing or interfere with the study conduct.
4. Subject has evidence of a systemic infection or has used systemic antibiotics for EB-related infections within 7 days before the screening visit (Visit 1).
5. Administration of systemic corticosteroids within 30 days (> 10 mg daily of prednisolone or corresponding) or of topical corticosteroids on target wound areas (primary, secondary and reference wound areas) within 14 days before the screening visit (Visit 1). Corticosteroids for inhalation, ophthalmic, or intranasal use are permitted.
6. Subject has undergone stem cell transplant or gene therapy for the treatment of EB with an effect on target wounds.
7. History of malignancy, including basal cell carcinomas or squamous cell carcinomas in the wound areas that will be included in the study.
8. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to TCP-25 or to any excipients of the hydrogel.
9. Planned treatment or treatment with another investigational drug within 3 months prior to Day -1.
10. Involvement in the planning and/or conduct of the study.
11. Investigator considers the patient unlikely to comply with study procedures, restrictions and requirements.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 15 days in Part I (modified endpoints & timeframes in Part II & III)
  Frequency, intensity and seriousness of adverse events (AEs)
Incidence of abnormal local reactions (Local tolerability) | Day 1 in Part I (modified endpoints & timeframes in Part II & III)
  Incidence of abnormal local reactions as compared to expected wound healing outcome, by direct assessment by Investigator:
  * Skin and wound erythema (abnormal reaction noted)
  * Skin and wound oedema and swelling (abnormal reaction noted)
  * Wound necrosis, crusting, and hemorrhage (abnormal reactions noted)
  * Wound purulent discharge as sign of excessive bacterial colonization and/or infection
Incidence of abnormal local reactions (Local tolerability) | Day 2 in Part I (modified endpoints & timeframes in Part II & III)
  Incidence of abnormal local reactions as compared to expected wound healing outcome, by direct assessment by Investigator:
  * Skin and wound erythema (abnormal reaction noted)
  * Skin and wound oedema and swelling (abnormal reaction noted)
  * Wound necrosis, crusting, and hemorrhage (abnormal reactions noted)
  * Wound purulent discharge as sign of excessive bacterial colonization and/or infection
Incidence of abnormal local reactions (Local tolerability) | Day 3 in Part I (modified endpoints & timeframes in Part II & III)
  Incidence of abnormal local reactions as compared to expected wound healing outcome, by direct assessment by Investigator:
  * Skin and wound erythema (abnormal reaction noted)
  * Skin and wound oedema and swelling (abnormal reaction noted)
  * Wound necrosis, crusting, and hemorrhage (abnormal reactions noted)
  * Wound purulent discharge as sign of excessive bacterial colonization and/or infection
Incidence of abnormal local reactions (Local tolerability) | Day 5 in Part I (modified endpoints & timeframes in Part II & III)
  Incidence of abnormal local reactions as compared to expected wound healing outcome, by direct assessment by Investigator:
  * Skin and wound erythema (abnormal reaction noted)
  * Skin and wound oedema and swelling (abnormal reaction noted)
  * Wound necrosis, crusting, and hemorrhage (abnormal reactions noted)
  * Wound purulent discharge as sign of excessive bacterial colonization and/or infection
Incidence of abnormal local reactions (Local tolerability) | Day 8 in Part I (modified endpoints & timeframes in Part II & III)
  Incidence of abnormal local reactions as compared to expected wound healing outcome, by direct assessment by Investigator:
  * Skin and wound erythema (abnormal reaction noted)
  * Skin and wound oedema and swelling (abnormal reaction noted)
  * Wound necrosis, crusting, and hemorrhage (abnormal reactions noted)
  * Wound purulent discharge as sign of excessive bacterial colonization and/or infection
Incidence of abnormal local reactions (Local tolerability) | Day 11 in Part I (modified endpoints & timeframes in Part II & III)
  Incidence of abnormal local reactions as compared to expected wound healing outcome, by direct assessment by Investigator:
  * Skin and wound erythema (abnormal reaction noted)
  * Skin and wound oedema and swelling (abnormal reaction noted)
  * Wound necrosis, crusting, and hemorrhage (abnormal reactions noted)
  * Wound purulent discharge as sign of excessive bacterial colonization and/or infection
Incidence of abnormal local reactions (Local tolerability) | Day 15 in Part I (modified endpoints & timeframes in Part II & III)
  Incidence of abnormal local reactions as compared to expected wound healing outcome, by direct assessment by Investigator:
  * Skin and wound erythema (abnormal reaction noted)
  * Skin and wound oedema and swelling (abnormal reaction noted)
  * Wound necrosis, crusting, and hemorrhage (abnormal reactions noted)
  * Wound purulent discharge as sign of excessive bacterial colonization and/or infection
Number of patients with clinically significant changes from baseline in electrocardiogram (ECG) | During screening (baseline) and on day 11 in Part I (modified endpoints & timeframes in Part II & III)
  Systolic and diastolic blood pressure and pulse will be measured. Any abnormalities will be specified and documented as clinically significant or not clinically significant by the investigator.
Number of patients with clinically significant changes from baseline in vital signs. | During screening (baseline) and on day 11 in Part I (modified endpoints & timeframes in Part II & III)
  Vital signs include systolic/diastolic blood pressure and pulse rate. Any vital signs outside the normal ranges will be judged as not clinically significant or clinically significant by the investigator.
Number of patients with clinically significant changes from baseline in physical examinations | During screening (baseline) and on day 11 in Part I (modified endpoints & timeframes in Part II & III)
  A physical examination will include assessments of general condition, lymph nodes, throat, heart, lungs and abdomen. Any abnormalities will be specified and documented as clinically significant or not clinically significant by the investigator.
Number of patients with clinically significant changes from baseline in safety laboratory parameters | During screening (baseline) and on day 2 in Part I (modified endpoints & timeframes in Part II & III)
  Safety laboratory parameters include haematology, clinical chemistry and coagulation. Any lab values outside the normal ranges will be judged as not clinically significant or clinically significant by the investigator.
  Haematology parameters to be measured are:
  * Haematocrit
  * Haemoglobin
  * Erythrocytes
  * Mean corpuscular volume
  * Mean corpuscular haemoglobin
  * Mean corpuscular haemoglobin concentration
  * Thrombocytes
  * Leukocytes
  * Eosinophils
  * Neutrophils
  * Basophils
  * Lymphocytes
  * Monocytes
  Clinical chemistry parameters to be measured are:
  * Alanine aminotransferase (ALT)
  * Aspartate aminotransferase (AST)
  * Creatinine
  * C-reactive protein (CRP)
  * Glucose
  * Haemoglobin A1c (HbA1C)
  Coagulation parameters to be measured are:
  * Activated partial thromboplastin time (APTT)
  * Prothrombin complex/International Normalised Ratio (PK/INR)
Number of patients with clinically significant changes from baseline in safety laboratory parameters | During screening (baseline) and on day 3 in Part I (modified endpoints & timeframes in Part II & III)
  Safety laboratory parameters include haematology, clinical chemistry and coagulation. Any lab values outside the normal ranges will be judged as not clinically significant or clinically significant by the investigator.
  Haematology parameters to be measured are:
  * Haematocrit
  * Haemoglobin
  * Erythrocytes
  * Mean corpuscular volume
  * Mean corpuscular haemoglobin
  * Mean corpuscular haemoglobin concentration
  * Thrombocytes
  * Leukocytes
  * Eosinophils
  * Neutrophils
  * Basophils
  * Lymphocytes
  * Monocytes
  Clinical chemistry parameters to be measured are:
  * Alanine aminotransferase (ALT)
  * Aspartate aminotransferase (AST)
  * Creatinine
  * C-reactive protein (CRP)
  * Glucose
  * Haemoglobin A1c (HbA1C)
  Coagulation parameters to be measured are:
  * Activated partial thromboplastin time (APTT)
  * Prothrombin complex/International Normalised Ratio (PK/INR)
Number of patients with clinically significant changes from baseline in safety laboratory parameters | During screening (baseline) and on day 5 in Part I (modified endpoints & timeframes in Part II & III)
  Safety laboratory parameters include haematology, clinical chemistry and coagulation. Any lab values outside the normal ranges will be judged as not clinically significant or clinically significant by the investigator.
  Haematology parameters to be measured are:
  * Haematocrit
  * Haemoglobin
  * Erythrocytes
  * Mean corpuscular volume
  * Mean corpuscular haemoglobin
  * Mean corpuscular haemoglobin concentration
  * Thrombocytes
  * Leukocytes
  * Eosinophils
  * Neutrophils
  * Basophils
  * Lymphocytes
  * Monocytes
  Clinical chemistry parameters to be measured are:
  * Alanine aminotransferase (ALT)
  * Aspartate aminotransferase (AST)
  * Creatinine
  * C-reactive protein (CRP)
  * Glucose
  * Haemoglobin A1c (HbA1C)
  Coagulation parameters to be measured are:
  * Activated partial thromboplastin time (APTT)
  * Prothrombin complex/International Normalised Ratio (PK/INR)
Number of patients with clinically significant changes from baseline in safety laboratory parameters | During screening (baseline) and on day 11 in Part I (modified endpoints & timeframes in Part II & III)
  Safety laboratory parameters include haematology, clinical chemistry and coagulation. Any lab values outside the normal ranges will be judged as not clinically significant or clinically significant by the investigator.
  Haematology parameters to be measured are:
  * Haematocrit
  * Haemoglobin
  * Erythrocytes
  * Mean corpuscular volume
  * Mean corpuscular haemoglobin
  * Mean corpuscular haemoglobin concentration
  * Thrombocytes
  * Leukocytes
  * Eosinophils
  * Neutrophils
  * Basophils
  * Lymphocytes
  * Monocytes
  Clinical chemistry parameters to be measured are:
  * Alanine aminotransferase (ALT)
  * Aspartate aminotransferase (AST)
  * Creatinine
  * C-reactive protein (CRP)
  * Glucose
  * Haemoglobin A1c (HbA1C)
  Coagulation parameters to be measured are:
  * Activated partial thromboplastin time (APTT)
  * Prothrombin complex/International Normalised Ratio (PK/INR)

SECONDARY OUTCOMES:
Plasma concentration of TCP-25 | Day 1 (measured before blister formation) in Part I (modified endpoints & timeframes in Part II & III)
  Measurement of TCP-25 concentration in plasma
Plasma concentration of TCP-25 | Day 2 (measured before administration of the intervention and 0.5 and 1 hours after administration of the intervention) in Part I (modified endpoints & timeframes in Part II & III)
  Measurement of TCP-25 concentration in plasma
Plasma concentration of TCP-25 | Day 3 (measured before administration of the intervention 1 hour after administration of the intervention) in Part I (modified endpoints & timeframes in Part II & III)
  Measurement of TCP-25 concentration in plasma
Plasma concentration of TCP-25 | Day 5 (measured before administration of intervention) in Part I (modified endpoints & timeframes in Part II & III)
  Measurement of TCP-25 concentration in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital in Lund, Clinical Trial Unit, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No
Publication of the study results and access to the study data is at the discretion of the Sponsor. It may be made available upon reasonable request.

REFERENCES:
- [Derived] Wallblom K, Forsberg F, Lundgren S, Fisher J, Cardoso J, Petruk G, Stromdahl AC, Saleh K, Puthia M, Schmidtchen A. Bactogram: Spatial Analysis of Bacterial Colonisation in Epidermal Wounds. Exp Dermatol. 2024 Dec;33(12):e70018. doi: 10.1111/exd.70018. PMID 39627888
- [Derived] Lundgren S, Wallblom K, Fisher J, Erdmann S, Schmidtchen A, Saleh K. Study protocol for a phase 1, randomised, double-blind, placebo-controlled study to investigate the safety, tolerability and pharmacokinetics of ascending topical doses of TCP-25 applied to epidermal suction blister wounds in healthy male and female volunteers. BMJ Open. 2023 Feb 22;13(2):e064866. doi: 10.1136/bmjopen-2022-064866. PMID 36813496